CLINICAL TRIAL: NCT03694080
Title: Calcium Electroporation for Early Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-188-2017
Record Dates: First submitted 2018-09-25; First posted 2018-10-03 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Calcium Electroporation treatment (Experimental): Calcium electroporation for colorectal cancer as a preoperative treatment before elective surgery.
  Interventions: Combination Product: Calcium electroporation

INTERVENTIONS:
Combination Product: Calcium electroporation — Patients with potentially curable colorectal rectal cancer will be treated preoperatively

SUMMARY:
This is an explorative, phase I clinical trial. The aim of this study is to establish the safety and efficacy of treating patients with early colorectal cancer with calcium electroporation prior to intended curative surgery.

DETAILED DESCRIPTION:
This is an explorative, phase I clinical trial. The aim of this study is to establish the safety and efficacy of treating patients with early colorectal cancer with calcium electroporation as a down staging and immune-response enhancing treatment prior to intended curative surgery. The study involves recruitment of patients with histologically verified rectal and sigmoid colon cancer with no indication for neoadjuvant chemoradiotherapy (experimental or standard care based) prior to intended curative surgery. In total the study will involve 24 patients, of these, 12 patients with rectal cancer and 12 patients with sigmoid colon cancer.

In relation to the intervention, clinical examination, blood samples, biopsies and questionnaires will be collected to evaluate safety, tumor respons and immunologic response to the treatment.

Patients will be followed for one month after the elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Patients must be mentally capable of understanding the information given.

  * Patients must give written informed consent.
  * Histologically verified adenocarcinoma of the rectum or sigmoid colon.
  * Tumor described as passable at index endoscopy.
  * Men or women aged at least 18 years.
  * Case reviewed by MDT (surgery, radiology, oncology). Case considered curable with standard surgical resection.
  * ASA class I-II (Classification of the American Society of Anesthesiology)

Exclusion Criteria:

* • Uncorrectable coagulation disorder.

  * Highly inflamed gastrointestinal tissue which is ulcerated and bleeding
  * Patients with ICD or pacemaker units.
  * Ongoing immunosuppressive treatment.
  * Patients with concomitant use of phenytoin.
  * Concurrent treatment with an investigational medicinal product.
  * Patients with any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study recruitments.
  * Advanced tumor stages, clinical UICC stage IV.
  * Indication for neoadjuvant chemoradiation or chemotherapy prior to surgery
  * Acute surgical resection.
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 42 days
  Safety will be evaluated through registration of adverse events related to the treatment. CTCAE will be used

SECONDARY OUTCOMES:
Histopathological characterization of the tumor | 14 days
  ypTNM staging and tumor regression grade according to current standards
Immunologic infiltration of the tumor tissue after calcium electroporation | 14 days
  Specific immunohistochemical staining for PD-1/PD-L1, CD3 and CD8 will be performed on biopsies and the final surgical specimen.
Immunoscore classification | 14 days
  Tumor infiltration on T-cells and subtypes will be characterized according to the immunoscore classification system.
Systemic immune response according to cytokine analysis | 42 days
  Blood samples will be collected prior to calcium electroporation and again at follow-up. Multiplex cytokine analysis will be performed
Systemic immune response according to flow cytometri | 42 days
  Blood samples will be collected prior to calcium electroporation and again at follow-up. Flow cytometri will be performed to evaluate immunological changes to the treatment.
Metastatic ability after potentially curable surgery | 42 days
  Cell adhesion assay will be performed on blood samples to evalutate the metastatic ability.
Cell proliferation as a marker for metastatic ability | 42 days
  Cell proliferation analyses will be performed on blood samples to evaluate metastatic ability

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, DMSc, Principal Investigator — Zealand University Hospital
Locations (1):
- Department of Surgery, Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: Undecided